CLINICAL TRIAL: NCT00918957
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center Phase III Study in Cystic Fibrosis (CF) Subjects to Assess Efficacy, Safety and Pharmacokinetics of Tobramycin Inhalation Powder From a Modified Manufacturing Process (TIPnew).
Brief Title: A Study of Tobramycin Inhalation Powder From a Modified Manufacturing Process Versus Placebo
Acronym: EDIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CTBM100C2303; 2008-002318-22 (EudraCT Number)
Record Dates: First submitted 2009-06-04; First posted 2009-06-11 (Estimated); Results first posted 2012-10-03 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-10

CONDITIONS: Cystic Fibrosis
Keywords: Tobramycin Inhalation Powder; Cystic fibrosis; Lung diseases; Anti-Bacterial Agents; Treatment of infections with P. aeruginosa in cystic fibrosis subjects
MeSH Terms: conditions — Cystic Fibrosis; Lung Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- TIP (Tobramycin Inhalation Powder) (Experimental): Tobramycin 28 mg powder. The TIP dose of 112 mg twice a day (bis in diem = b.i.d.), given in a cycle of 28 days on treatment followed by 28 days off treatment.
  Interventions: Drug: Tobramycin Inhalation Powder
- Placebo (Placebo Comparator): Placebo 20 mg powder capsules. The dose regimen for the reference product was inhaling the contents of four capsules twice a day (bis in diem = b.i.d.), in the morning and in the evening for 28 days (on treatment), followed by 28 days of no study treatment (off treatment).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tobramycin Inhalation Powder — Tobramycin Inhalation Powder as produced by a modified manufacturing process TIP. TIP was provided in hard capsules each containing 28 mg active ingredient (tobramycin); Capsules were packaged in blister cards and administered by the T-326 Inhaler.
  Arms: TIP (Tobramycin Inhalation Powder)
Drug: Placebo — Placebo inhalation powder consisting of the excipients used for TIP. Placebo was provided in hard capsules, containing 20 mg placebo powder, which were packaged in blister cards, matching in appearance to TIP. Capsules were administered by the T-326 Inhaler.
  Arms: Placebo

SUMMARY:
This study is designed to show how well tobramycin inhalation powder works and how safe it is when produced by a modified manufacturing process

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent given by adults or by the parents/legal guardian in combination with the patient's assent, if capable of assenting, before any assessment was performed
* Confirmed diagnosis of Cystic Fibrosis (CF) by the presence of one or more clinical features of CF in addition to:

  * a quantitative pilocarpine iontophoresis sweat chloride test of >60 mEq/L; or
  * identification of well-characterized disease-causing mutations in each CFTR gene; or
  * an abnormal nasal transepithelial potential difference characteristic of CF.
* Forced Expiratory Volume in one second (FEV1) at screening must have been ≥25% and ≤80% of normal predicted values for age, sex, and height based on Knudson criteria
* P. aeruginosa must have been present in a sputum/deep-throat cough swab culture (or bronchoalveolar lavage [BAL]) within 6 months prior to screening and in the sputum/deep-throat cough swab culture at the screening visit
* Able to expectorate a sputum sample or provide a deep throat cough swab at screening
* Able to comply with all protocol requirements
* Use of an effective means of contraception in females of childbearing potential
* Clinically stable in the opinion of the investigator to be treated according to this protocol

Exclusion Criteria:

* FEV1 at baseline (Visit 2) <25% or >80% of normal predicted values for age, sex, and height based on Knudson criteria, and/or FEV1 at baseline (Visit 2) deviated by ≥10% from the FEV1 measured at screening (Visit 1)
* Any use of inhaled anti-pseudomonal antibiotics within 4 months prior to screening
* Any use of systemic anti-pseudomonal antibiotics within 28 days prior to study drug administration
* Serum creatinine 2 mg/dL or above, blood urea nitrogen (BUN) 40 mg/dL or above, or an abnormal urinalysis defined as 2+ or greater proteinuria
* Known local or systemic hypersensitivity to aminoglycosides or inhaled antibiotics
* Signs and symptoms of acute pulmonary disease, e.g. pneumonia, pneumothorax
* Administration of any investigational drug within 30 days prior to enrollment
* Any previous exposure to tobramycin dry powder for inhalation (TIP)
* Administration of loop diuretics within 7 days prior to study drug administration
* Initiation of treatment with chronic macrolide therapy within 28 days prior to study drug administration
* Initiation of treatment with dornase alfa within 28 days prior to study drug administration
* Initiation of treatment with inhaled steroids (or increased dose) within 28 days prior to study drug administration
* Initiation of treatment with inhaled hypertonic saline (HS) within 28 days prior to study drug administration
* Personal history of abnormal hearing or family history of abnormal hearing other than typical hearing loss associated with the aging process
* Known abnormal result from any audiology testing (defined as either a unilateral puretone audiometry test showing a threshold elevation >20 dB at any frequency across the frequency range 0.25 kHz to 8 kHz or the absence of emission at the evoked otoacoustic emission test)
* History of sputum culture or throat swab (or BAL) culture yielding Burkholderia cepacia (B. cepacia) within 2 years prior to screening and/or sputum culture yielding B. cepacia at screening
* Hemoptysis of more than 60 mL at any time within 30 days prior to study drug administration
* History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of evidence of local recurrence or metastases
* Patients with clinically significant laboratory abnormalities (not associated with the study indication) at screening
* Patients or caregivers with a history of noncompliance to medical regimens and patients or caregivers who are considered potentially unreliable
* Pregnant or nursing (lactating) women
* Women of child-bearing potential unless they used two reliable birth control methods

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2009-06; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (24):
- Bulgaria (4):
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Varna
- Egypt (2):
  - Novartis Investigative Site, Alexandria
  - Novartis Investigative Site, Giza
- Estonia (2):
  - Novartis Investigative Site, Tallinn
  - Novartis Investigative Site, Tartu
- India (4):
  - Novartis Investigative Site, Chandigarh
  - Novartis Investigative Site, Hyderabad
  - Novartis Investigative Site, New Delhi
  - Novartis Investigative Site, Vellore
- Novartis Investigative Site, Riga, Latvia
- Lithuania (2):
  - Novartis Investigative Site, Kaunas
  - Novartis Investigative Site, Vilnius
- Romania (2):
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Timișoara
- Russia (6):
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Samara
  - Novartis Investigative Site, Voronezh
  - Novartis Investigator Site, Yaroslavi
- Novartis Investigative Site, Durban, South Africa

REFERENCES:
- [Derived] Galeva I, Konstan MW, Higgins M, Angyalosi G, Brockhaus F, Piggott S, Thomas K, Chuchalin AG. Tobramycin inhalation powder manufactured by improved process in cystic fibrosis: the randomized EDIT trial. Curr Med Res Opin. 2013 Aug;29(8):947-56. doi: 10.1185/03007995.2013.805122. Epub 2013 Jun 5. PMID 23672633

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Although 32 patients were randomized to the TIP group and 30 to the Placebo group, the ITT population included 2 patients allocated to the TIP group but received placebo due to Investigator error during the drug dispensation process. The safety population contained 30 patients who were treated with TIP and 32 patients who were treated with placebo.
Groups:
- Placebo: Placebo 20 mg powder capsules. The dose regimen for the reference product was inhaling the contents of four capsules twice a day (bis in diem = b.i.d.) in the morning and in the evening for 28 days (on treatment), followed by 28 days of no study treatment (off treatment).
Period: Overall Study
Arm/Group | TIP (Tobramycin Inhalation Powder) | Placebo
Started | 32 | 30
Completed | 29 | 30
Not Completed | 3 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TIP (Tobramycin Inhalation Powder) | Placebo | Total
Number analyzed (Participants) | 30 | 32 | 62
Age Continuous [Mean (Standard Deviation); unit: years] | 12.9 (4.25) | 12.9 (4.68) | 12.9 (4.44)
Age, Customized [Number; unit: participants]
  <13 years | 15 | 15 | 30
  >= 13 years | 15 | 17 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 19 | 40
  Male | 9 | 13 | 22
Baseline Forced Expiratory Volume in one second (FEV1) percentage predicted [Mean (Standard Deviation); unit: Percentage] — * Any spirometry values that are listed as missing at Screening and/or Baseline FEV1 % predicted can include data that was captured but identified as technically unacceptable.
  * Baseline is defined as the latest measurement prior to first dosing of study medication.
  Percentage | 59.1 (18.18) | 59.3 (16.61) | 59.2 (17.25)
Baseline P. aeruginosa sputum density [Mean (Standard Deviation); unit: Log10 CFU (colony forming unit)] — * Overall density, defined as the sum of biotypes (mucoid, dry and small colony variant).
  * Baseline is defined as the latest measurement prior to first dosing of study medication.
    * If sub-isolates existed for CFU biotype mucoid or dry, then the sum of sub-isolates is analyzed.
  Log10 CFU (colony forming unit) | 7.4 (1.53) | 7.4 (1.55) | 7.4 (1.52)

OUTCOME MEASURES:

1. Primary Outcome: Relative Change From Baseline of Forced Expiratory Volume in One Second (FEV1) Percent Predicted to End of Dosing (Day 29)
Description: Relative change in percentage predicted FEV1 in the Intent-to-treat (ITT), modified ITT (mITT) and Observed cases in the ITT populations were calculated from an adjusted analysis ANOVA model.
  ITT Patients with missing or unacceptable Day 29 spirometry measurements had their primary endpoint data imputed with zero.
  BSL = Baseline, defined as the latest measurement prior to the first dosing of study medication
  - Relative change = 100 * (value - baseline) / baseline There were 3 patients who had no screening nor baseline values (due to inadequate spirometry) and so were excluded from all change from baseline analyses.
Time Frame: Baseline, Day 29
Population: ITT: All randomized patients (pts) received at least one dose of study drug. Missing or unacceptable Day 29 spirometry test -change from baseline FEV1 % predicted imputed using last available post-baseline value or 0. mITT: Pts with unacceptable FEV1 measurements excluded. Observed cases: Pts with missing or unacceptable FEV1 measurements excluded.
Measure: Least Squares Mean (Standard Error); unit: change in percentage
Arm/Group | TIP (Tobramycin Inhalation Powder) | Placebo
Number analyzed (Participants) | 31 | 28
change in percentage
  Participants analyzed: ITT Population (31, 28) | 8.2 (2.93) [2.3 to 14.1] | 2.3 (3.13) [-4.0 to 8.6]
  Parts. analyzed: Modified ITT Pop (27, 27) | 9.7 (3.30) [3.1 to 16.3] | 2.5 (3.30) [-4.1 to 9.2]
  Parts analyzed: Observed Cases in ITT Pop (25, 27) | 10.3 (3.42) [3.4 to 17.2] | 2.4 (3.35) [-4.3 to 9.2]

2. Secondary Outcome: Change From Baseline of Forced Vital Capacity (FVC) Percent Predicted to End of Dosing (Day 29) and to the End of Off-cycle Period (Day 57)
Description: Results of statistical analysis were calculated from an ANOVA model. Baseline is defined as the latest measurement prior to the first dosing of study medication.
  Response (percentage change) = treatment + Screening FEV1 percentage predicted (<50 and >=50) + age (<13 and >=13) + error
Time Frame: Baseline, Day 29, Day 57
Population: Intent-to-treat (ITT) population: All randomized patients who received at least one dose of study drug. Following the intent-to-treat principle, patients were analyzed according to the treatment they were assigned to at randomization.
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | TIP (Tobramycin Inhalation Powder) | Placebo
Number analyzed (Participants) | 31 | 28
percentage change
  Number of participants analyzed (31, 28): Baseline | 73.3 (19.19) | 76.9 (15.16)
  Number of participants analyzed (25, 27): Day 29 | 7.2 (9.94) [1.1 to 10.4] | 1.6 (14.74) [-3.4 to 6.6]
  Number of participants analyzed (28, 23): Day 57 | 5.2 (16.99) | 3.1 (15.05)

3. Secondary Outcome: Change From Baseline of Forced Expiratory Flow Rate Over 25 and 75 Percent. (FEF25-75%) Predicted to End of Dosing (Day 29) and End of Off-cycle Period (Day 57)
Description: FEF25-75: Forced expiratory flow rate over 25% to 75% of vital capacity
  For FEF25-75 percentage predicted the relative change is analyzed. If screening FEV1 percentage predicted is missing, it will be imputed by the baseline value.
Time Frame: Baseline, Day 29, Day 57
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | TIP (Tobramycin Inhalation Powder) | Placebo
Number analyzed (Participants) | 31 | 28
percentage change
  Number of participants analyzed (31, 28): Baseline | 36.2 (20.15) | 35.9 (20.67)
  Number of participants analyzed (25, 27): Day 29 | 21.00 (36.55) [4.7 to 28.3] | 7.8 (29.65) [-5.9 to 19.3]
  Number of participants analyzed (28, 23): Day 57 | 23.9 (35.57) | 17.7 (37.40)

4. Secondary Outcome: Absolute Change From Baseline to End of Dosing (Day 29) and End of Off-cycle Period (Day 57) in Sputum Pseudomonas Aeruginosa Density (log10 Colony Forming Units(CFU) Per Gram Sputum)
Description: P. aeruginosa sputum density refers to overall density, defined as the sum of biotypes (mucoid, dry and small colony variant).
  If sub-isolates exist for CFU biotype mucoid or dry, then the sum of sub-isolates is analyzed.
Time Frame: Baseline, Day 29, Day 57
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Log10 CFU (colony forming unit)
Arm/Group | TIP (Tobramycin Inhalation Powder) | Placebo
Number analyzed (Participants) | 31 | 28
Log10 CFU (colony forming unit)
  Number of participants analyzed (29, 28): Baseline | 7.5 (1.49) | 7.3 (1.58)
  Number of participants analyzed (14, 27): Day 29 | -2.4 (1.54) [-1.7 to -0.7] | 0.0 (0.89) [-0.6 to 0.5]
  Number of participants analyzed (19, 24): Day 57 | -0.9 (2.09) | -0.2 (1.20)

5. Secondary Outcome: Change From Baseline to End of Dosing (Day 29) and End of Off-cycle Period (Day 57) of Pseudomonas Aeruginosa Minimum Inhibitory Concentration (MIC)
Description: Maximum MIC values from all biotypes were used. Absolute values and changes in tobramycin MIC for P. aeruginosa from baseline are summarized by biotype. Overall, a high variability of MIC was observed within each treatment group. For the maximum of all biotypes, large differences in mean changes from baseline at Day 29 were observed between the TIP group and the placebo group.
Time Frame: Baseline, Day 29, Day 57
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | TIP (Tobramycin Inhalation Powder) | Placebo
Number analyzed (Participants) | 31 | 28
μg/mL
  Number of participants analyzed (28, 29):Baseline | 0.8 (1.49) | 2.7 (11.81)
  Number of participants analyzed (13, 27): Day 29 | 0.1 (0.73) | 10.0 (38.32)
  Number of participants analyzed (19, 24): Day 57 | 0.5 (1.49) | 1.4 (6.58)

6. Secondary Outcome: Shift From Baseline in Laboratory Parameters to Above Upper/Lower Limit of Normal
Description: Hematology values shift from baseline to above upper/below lower limit of normal at any time post-baseline.
  Biochemistry values shift from baseline to above upper/below lower limit of normal at any time post-baseline.
Time Frame: Baseline, Study completion
Population: Safety population: All randomized patients who received at least one dose of study drug. In all safety analyses patients were analyzed according to the treatment received.
Measure: Number; unit: percentage of participants at risk
Arm/Group | TIP (Tobramycin Inhalation Powder) | Placebo
Number analyzed (Participants) | 30 | 32
percentage of participants at risk
  Hematology (Hem): Absolute Basophilis- low - low | 0.0 | 0.0
  Hem: Absolute Basophilis - high | 8.3 | 10.0
  Hem: Absolute Eosinophils - low | 0.0 | 0.0
  Hem: Absolute Eosinophils - high | 14.3 | 7.4
  Hem: Absolute Lymphocytes - low | 4.2 | 3.7
  Hem: Absolute Lymphocytes - high | 11.1 | 9.5
  Hem: Absolute Monocytes - low | 0.0 | 0.0
  Hem: Absolute Monocytes - high | 9.5 | 19.2
  Hem: Absolute Neutrophils (Seg. + Bands) - low | 9.5 | 10.3
  Hem: Absolute Neutrophils (Seg. + Bands) - high | 11.1 | 25.0
  Hem: Basophils - low | 0.0 | 0.0
  Hem: Basophils - high | 60.0 | 40.0
  Hem: Eosinophils - low | 0.0 | 0.0
  Hem: Eosinophils - high | 28.6 | 14.8
  Hem: Lymphocytes -low | 4.3 | 14.3
  Hem: Lymphocytes - high | 14.3 | 7.7
  Hem: Monocytes - low | 8.3 | 0.0
  Hem: Monocytes - high | 27.8 | 24.0
  Hem: Neutrophils (Seg. + Bands) - low | 13.6 | 11.1
  Hem: Neutrophils (Seg. + Bands) - high | 4.3 | 6.9
  Hem: Platelet count (direct) - low | 4.5 | 0.0
  Hem: Platelet count (direct) - high | 7.7 | 13.3
  Hem: RBC- low | 0.0 | 0.0
  Hem: RBC- high | 16.7 | 9.1
  Hem: WBC (total)- low | 9.5 | 3.7
  Hem: WBC (total) - high | 5.3 | 26.1
  Hem: Hematocrit - low | 0.0 | 0.0
  Hem: Hematocrit - high | 14.3 | 14.8
  Hem: Hemoglobin - low | 3.8 | 0.0
  Hem: Hemoglobin - high | 4.2 | 3.3
  Biochemistry (Bio): Album - low | 0.0 | 0.0
  Bio: Album - high | 20.0 | 10.0
  Bio: Alkaline phosphatase, serum - low | 0.0 | 0.0
  Bio: Alkaline phosphatase, serum - high | 14.3 | 4.3
  Bio: Bilirubin (direct/conjugated) -low | 0.0 | 0.0
  Bio: Bilirubin (direct/conjugated) -high | 7.7 | 7.1
  Bio: Bilirubin (total) - low | 0.0 | 0.0
  Bio: Bilirubin (total) - high | 3.4 | 3.3
  Bio: Blood Urea Nitrogen (BUN) - low | 0.0 | 13.8
  Bio: Blood Urea Nitrogen (BUN) - high | 3.4 | 3.2
  Bio: Calcium -low | 0.0 | 12.9
  Bio: Calcium -high | 6.9 | 6.7
  Bio: Chloride - low | 0.0 | 6.5
  Bio: Chloride - high | 10.3 | 0.0
  Bio: Creatinine - low | 0.0 | 50.0
  Bio: Creatinine - high | 0.0 | 0.0
  Bio: Gamma Glutamyltransferase - low | 0.0 | 3.2
  Bio: Gamma Glutamyltransferase - high | 4.2 | 3.8
  Bio: Glucose - low | 12.0 | 20.0
  Bio: Glucose - high | 11.1 | 6.7
  Bio: Phosphate (Inorganic Phosphorus) - low | 0.0 | 0.0
  Bio: Phosphate (Inorganic Phosphorus) - high | 19.2 | 13.8
  Bio: Potassioum - low | 0.0 | 3.2
  Bio: Potassioum - high | 7.1 | 0.0
  Bio: SGOT (AST) - low | 0.0 | 3.2
  Bio: SGOT (AST) - high | 12.5 | 12.0
  Bio: SGPT (ALT) - low | 0.0 | 0.0
  Bio: SGPT (ALT) - high | 9.5 | 13.0
  Bio: Serum bicarbonate - low | 47.6 | 23.8
  Bio: Serum bicarbonate - high | 0.0 | 0.0
  Bio: Sodium - low | 0.0 | 6.5
  Bio: Sodium - high | 10.3 | 0.0
  Bio: Total Protein (Serum) - low | 0.0 | 3.2
  Bio: Total Protein (Serum) - high | 4.2 | 29.2
  Bio: Uric Acid - low | 3.6 | 3.2
  Bio: Uric Acid - high | 10.7 | 19.2

7. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: Adverse Events (AEs) (on and off treatment) regardless of study relationship by primary system organ and treatment group.
  Primary system organ classes are sorted in descending order of frequency in the TIP treatment group.
  A patient with more than one AE within a primary system organ class is counted only once for that class.
Time Frame: First administration of study drug, study completion
Population: Safety population: All randomized patients who received at least one dose of study drug.In all safety analyses patients were analyzed according to the treatment received
Measure: Number; unit: Percentage of participants
Arm/Group | TIP (Tobramycin Inhalation Powder) | Placebo
Number analyzed (Participants) | 30 | 32
Percentage of participants
  Respiratory, thoracic & mediastinal disorders | 13.3 | 3.1
  Ear and labyrinth disorders | 10.0 | 6.3
  Infections and infestations | 10.0 | 25.0
  Gastrointestinal disorders | 3.3 | 3.1
  Metabolism and nutrition disorders | 3.3 | 3.1
  Nervous system disorders | 3.3 | 0.0
  Renal and urinary disorders | 3.3 | 0.0
  Skin and subcutaneous tissue disorder | 3.3 | 0.0
  Blood and lymphatic system disorder | 0.0 | 3.1
  Injury, poisoning and procedural complications | 0.0 | 3.1
  Investigation | 0.0 | 3.1

8. Secondary Outcome: Percentage of Participants With Serious Adverse Events (SAEs)
Description: Serious Adverse Events (on and off treatment) by preferred term and treatment group.
  Preferred terms are sorted in descending order of frequency in the TIP treatment group.
  A patient with multiple occurrences of the same preferred term is counted only once in the preferred term.
Time Frame: Time of consent, 4 weeks after study completion
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | TIP (Tobramycin Inhalation Powder) | Placebo
Number analyzed (Participants) | 30 | 32
percentage of participants
  Lower limb fracture | 0.0 | 3.1
  Pneumonia | 0.0 | 3.1

9. Secondary Outcome: Acute Change in Airways Reactivity (FEV1 Percent Predicted) From Pre-dose to 30 Minutes After Completion of First Dose of Study Drug
Description: Relative change = 100 * (30-m-post-dose - pre-dose)/pre-dose assessed by the number and percentage of patients with a decrease of ≥20 % in FEV1 % predicted from pre dose to 30 minutes post dose.
  Day 1 is the scheduled visit of first study drug administration.
Time Frame: Day 1, Day 29
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | TIP (Tobramycin Inhalation Powder) | Placebo
Number analyzed (Participants) | 30 | 32
Percentage of participants
  Day 1 | 4.8 | 0.0
  Day 29 | 0.0 | 8.0

10. Secondary Outcome: Tobramycin Serum Concentration
Description: Descriptive statistics of serum and sputum concentrations per scheduled sampling time.
  Detectable concentration values at pre-dose on Day 1 were excluded from the analysis.
Time Frame: Pre-dose, 0 - 1 hour post-dose, 1 -2 hours post-dose, 2 - 6 hours post-dose
Population: Safety population: All randomized patients who received at least one dose of study drug. In all safety analyses patients were analyzed according to the treatment received.
  This measures the concentration of active substance in the body at different time-point to evaluate there is abnormal accumulation of active substance. Not for Placebo Patients.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | TIP (Tobramycin Inhalation Powder)
Number analyzed (Participants) | 30
μg/mL
  Day1: 0 -1 hour (hr) post dose (28, 0) | 0.83 (0.40)
  Day 1: 1 -2 hours (hr) post dose (28, 0) | 0.93 (0.44)
  Day 1: 2 -6 hours (hr) post dose (29, 0) | 0.73 (0.39)
  Day 29: Pre-dose (27, 0) | 0.41 (0.51)
  Day 29: 0 -1 hr post dose (28, 0) | 1.48 (0.69)
  Day 29: 1 -2 hrs post dose (29, 0) | 1.37 (0.64)
  Day 29: 2 -6 hrs post dose (27, 0) | 1.14 (0.65)

11. Primary Outcome: Pre-planned Sensitivity Analysis: Absolute Change From Baseline of Forced Expiratory Volume in One Second (FEV1) Percent (%) Predicted to End of Dosing (Day 29)
Description: Absolute change in percentage predicted FEV1 in the Intent-to-treat (ITT), modified ITT (mITT) and Observed cases in the ITT populations were calculated from an adjusted analysis ANOVA model.
  In the adjusted analysis model: response = treatment + screening FEV1 % predicted (<50 and >=50) + age (<13 and >=13) + error.
  Significance for the FEV1 % predicted is reached for p-values <= 0.05. There were 3 patients who had no screening nor baseline values (due to inadequate spirometry) and so were excluded from all change from baseline analyses.
Time Frame: Baseline, Day 29
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: change in percentage
Arm/Group | TIP (Tobramycin Inhalation Powder) | Placebo
Number analyzed (Participants) | 31 | 28
change in percentage
  Participants analyzed: ITT Population (31, 28) | 4.9 (1.59) | 0.5 (1.70)
  Parts. analyzed: Modified ITT Pop (25, 27) | 5.7 (1.78) | 0.6 (1.79)
  Parts. analyzed: Observed Cases, ITT Pop (27, 27) | 6.1 (1.84) | 0.5 (1.80)

12. Primary Outcome: Post-hoc: Relative Change From Baseline of Forced Expiratory Volume in One Second (FEV1) Percent Predicted to End of Dosing (Day 29) Without Outlier
Description: Relative change in percentage predicted FEV1 without outlier (outliers with respect to FEV1 values and PK data), in the Intent-to-treat (ITT), modified ITT (mITT) and Observed cases in the ITT populations were calculated from an adjusted analysis ANOVA model.
Time Frame: Baseline, Day 29
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: change in percentage
Arm/Group | TIP (Tobramycin Inhalation Powder) | Placebo
Number analyzed (Participants) | 31 | 28
change in percentage
  Participants analyzed: ITT Population (30, 28) | 10.4 (2.81) | 3.1 (2.92)
  Parts. analyzed: Modified ITT Pop (24, 27) | 12.4 (3.14) | 3.5 (3.05)
  Parts. analyzed: Observed Cases, ITT Pop (26, 27) | 13.1 (3.25) | 3.4 (3.08)

ADVERSE EVENTS:
Arm/Group | TIP (Tobramycin Inhalation Powder) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/30 | 2/32
Other Adverse Events (participants affected / at risk) | 4/30 | 6/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TIP (Tobramycin Inhalation Powder) (N=30) | Placebo (N=32)
Pneumonia (Infections and infestations) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TIP (Tobramycin Inhalation Powder) (N=30) | Placebo (N=32)
Hypoacusis (Ear and labyrinth disorders) | 3 | 2
Respiratory tract infection (Infections and infestations) | 0 | 2
Respiratory tract infection viral (Infections and infestations) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.